CLINICAL TRIAL: NCT04423965
Title: A Multicenter Randomized Controlled Phase II Trial of Neoadjuvant mFOLFOXIRI Versus Routine Chemoradiotherapy in the EMVI Positive Locally Advanced Rectal Cancer (TRICHEMO)
Brief Title: A Trial of Neoadjuvant mFOLFOXIRI Versus CRT in the EMVI Positive LARC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Collaborators: First Affiliated Hospital of Wenzhou Medical University (Other); Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Guosheng Wu, Chief physician, First Affiliated Hospital of Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TRICHEMO
Record Dates: First submitted 2020-06-08; First posted 2020-06-09 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Locally Advanced Rectal Cancer
MeSH Terms: interventions — Chemoradiotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- mFOLFOXIRI (Experimental): Patients receive 6 cycles of mFOLFOXIRI
  Interventions: Drug: mFOLFOXIRI
- Chemoradiotherapy(CRT) (Experimental): Patients receive standard chemoradiotherapy
  Interventions: Combination Product: Chemoradiotherapy

INTERVENTIONS:
Drug: mFOLFOXIRI — irinotecan 165 mg/m² IV day 1+ oxaliplatin 85 mg/m² IV day 1 + leucovorin 400 mg/m² day 1, fluorouracil 1200mg/m²/day *2 days (total 2400 mg/m² over 48 hours) continuous infusion starting on day 1 of each 2 weeks cycle
  Arms: mFOLFOXIRI
Combination Product: Chemoradiotherapy — Capecitabine based chemoradiotherapy
  Arms: Chemoradiotherapy(CRT)

SUMMARY:
Extramural Vascular Invasion Positive(EMVI+) is a high risk of distant metastasis for locally advanced rectal cancer(LARC) after resection. The study is to evaluate the efficacy and safety of FOLFOXIRI as neoadjuvant chemotherapy alone for EMVI+ LARC in contrast to the efficacy of standard Chemoradiotherapy (CRT).

DETAILED DESCRIPTION:
It is an investigator-initiated, multicentered, randomized controlled clinical study to evaluate the efficacy and safety of mFOLFOXIRI as neoadjuvant chemotherapy alone for EMVI+ LARC in contrast to standard chemoradiotherapy. Patients of LARC with EMVI+ evaluated by pelvic magnetic resonance imaging (MRI) are enrolled in this trial. All patients will be randomized divided into two groups.

Experimental group will receive 3 cycles of mFOLFOXIRI, followed to be performed MRI to assess clinical response. If the tumor response is good enough (partial response or complete response), the patient will receive another 3 cycles of mFOLFOXIRI then surgery. On the contrary, if the tumor shows poor response (stable disease or progressive disease) or with mesorectal fascia-positive or ycT4a/b after re-evaluation, radiotherapy will be performed combined with capecitabine before operation. Control group will receive standard capecitabine based chemoradiotherapy.

Patients with mesorectal fascia-positive or ycT4a/b after re-evaluation would receive radiation before surgery, whereas responders would have immediate total mesorectal excision (TME). All patients will receive 4 cycles of XELOX as adjuvant chemotherapy after TME.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥ 18 to 70 years at diagnosis;
2. ECOG status 0-2;
3. Diagnosis of rectal adenocarcinoma(Distal border of the tumor must be located < 12 cm from the anal verge);
4. MRI examination diagnosed EMVI-positive;
5. Tumor amenable to curative resection;
6. Adequate bone marrow, hepatic and renal function as assessed by the following laboratory requirements conducted within 7 days of starting study treatment: (1) Neutrophilic granulocytes ≥ 3.0 x10^9/L, Platelet count ≥ 75 x 10^9/L, Hemoglobin (Hb) ≥ 90g/L; (2) bilirubin ≤1.5 x the upper limit of normal (ULN),Alanine aminotransferase (ALT)/Aspartate aminotransferase (AST) ≤ 2.5 x ULN; (3) Serum creatinine ≤ 1.5 x ULN.No renal disease that would preclude study treatment or follow-up
7. Signed informed consent; able to comply with study and/or follow- up procedures

Exclusion Criteria:

1. Hypersensitivity to fluorouracil, oxaliplatin or irinotecan;
2. Patient had received pelvic radiotherapy;
3. Patient had received systemic chemotherapy;
4. History of invasive colon or rectal malignancy, regardless of disease-free interval;
5. Had metastatic disease;
6. Patient had second malignant disease within 5 years;
7. Uncontrolled co-morbid illnesses or other concurrent disease;
8. Patients refused to signed informed consent.
9. Pregnant and Nursing women

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2020-05-12 (Actual); Primary Completion 2022-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
MFS | 3 years
  metastasis free survival

SECONDARY OUTCOMES:
Tumor downstaging rate | 2 years
  the proportion of tumor downstaging to ypT0-2N0M0
pCR | 2 years
  Pathologic complete response rate
RFS | 3 years
  recurrence-free survival
DFS | 3 years
  disease-free survival
OS | 5 years
  overall survival
Reported Adverse events | 2 years
  The incidence of >=3 grade adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No